CLINICAL TRIAL: NCT05833802
Title: A Companion Trial in Silico: Computing Drug Response for Cancer Patients in Clinical Trials（PRincipal-001)
Brief Title: Computation Prediction of Drug Response Based on Omics Data
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Beijing Phil Rivers Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022YJZ109
Record Dates: First submitted 2023-03-24; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: in silico clinical trial; anti-cancer drug
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Screening Assays, Antitumor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- the virtual cohort: the virtual cohort that enroll in silico clinical trial (ISCT), and will be treated by virtual anti-cancer drug.
  Interventions: Other: virtual anti-cancer drug
- the real cohort: the real cohort that enroll in real word study, and will be treated by anti-cancer drug.

INTERVENTIONS:
Other: virtual anti-cancer drug — the virtual anti-cancer drug was formulation generated by computer modeling and artificial intelligence technology
  Other Names: anti-cancer drug
  Groups: the virtual cohort

SUMMARY:
The goal of this observational study is to assess the performance of computational medicine technology in predicting patients response to anticancer drugs based on omics data.The main question it aims to answer is test consistency between the computing drug response and the response of real-world clinical trials. Participants will take part in silico.

DETAILED DESCRIPTION:
A companion trial in silico was planned to compare head-to-head with a real clinical study of anti-tumor registered new drugs to verify the consistency between the efficacy prediction results of virtual clinical studies and the efficacy results of traditional clinical trials.

Subjects simultaneously entered real world clinical trials and virtual clinical trials built by computer modeling and artificial intelligence technology. The results of traditional clinical trials were compared with those of virtual clinical trials to calculate the consistency of virtual clinical trials.

By predicting the population with consistent efficacy, locking the response population to new drugs, using the innovative technology of computational medicine, grasping the omics characteristics of the response population, and using this as a starting point to determine the target population of clinical trials, so as to determine new screening conditions, design new clinical trials, accurately match the effective population, and revolutionary change the efficiency of clinical trials, thereby shortening the process and cost of clinical trial development.

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of triple-negative breast cancer
2. The subjects agreed to participate in the traditional clinical trial and signed informed consent.
3. The subjects agreed to participate in the virtual study and signed informed consent.

Exclusion Criteria:

1. Subjects do not meet the inclusion criteria of traditional clinical trial.
2. Subjects suffered from other cancer disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients with triple-negative breast cancer will participate in the traditional clinical trials and be treated by anti-cancer drug.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
consistency | 8 weeks after the first administration of the drug for subjects
  To compare the consistency of the tumor response between two cohorts. Tumor response for Patients in traditional clinical trial cohort will be assessed by New response evaluation criteria in solid tumours v1.1. Tumor response for virtual patients in virtual study will be predicted by the trained model.The efficacy prediction model will be trained using 4-5 patients evaluated for tumor response according to New response evaluation criteria in solid tumours v1.1, including at least 2 patients with Complete Response or Partial Response . The training of this model is based on the Damage Assessment of Genomic Mutations algorithm（EBioMedicine. 2021 Jul;69:103446）with the input of patients' genomic data.

CONTACTS AND LOCATIONS:
Overall Officials: Min Jiang, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Shuhua Zhao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olivier M, Asmis R, Hawkins GA, Howard TD, Cox LA. The Need for Multi-Omics Biomarker Signatures in Precision Medicine. Int J Mol Sci. 2019 Sep 26;20(19):4781. doi: 10.3390/ijms20194781. PMID 31561483
- [Background] Yang M, Fan Y, Wu ZY, Gu J, Feng Z, Zhang Q, Han S, Zhang Z, Li X, Hsueh YC, Ni Y, Li X, Li J, Hu M, Li W, Gao H, Yang C, Zhang C, Zhang L, Zhu T, Cheng M, Ji F, Xu J, Cui H, Tan G, Zhang MQ, Liang C, Liu Z, Song YQ, Niu G, Wang K. DAGM: A novel modelling framework to assess the risk of HER2-negative breast cancer based on germline rare coding mutations. EBioMedicine. 2021 Jul;69:103446. doi: 10.1016/j.ebiom.2021.103446. Epub 2021 Jun 19. PMID 34157485
- [Background] DiMasi JA, Grabowski HG, Hansen RW. Innovation in the pharmaceutical industry: New estimates of R&D costs. J Health Econ. 2016 May;47:20-33. doi: 10.1016/j.jhealeco.2016.01.012. Epub 2016 Feb 12. PMID 26928437
- See also: The latest global cancer burden data for 2020 — https://gco.iarc.fr/
- See also: Annual progress report on clinical trials of new drug registration in China ( 2021 ) — https://www.cde.org.cn/main/news/viewInfoCommon/1839a2c931e1ed43eb4cc7049e189cb0
- See also: At the end of 2021, Center for Drug Evaluation of National Medical Products Administration issued the Guideline: Guiding principles for clinical research and development of anti-tumor drugs ' — https://www.cde.org.cn/zdyz/domesticinfopage?zdyzIdCODE=67c30813bd94792b5b2a9f9bd7121763